CLINICAL TRIAL: NCT03546036
Title: Kontrollerad Studie av Behandling Med kedjetäcken Mot sömnstörning
Brief Title: Controlled Study of Chain Blanket for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Mats Adler, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/102-31/2
Record Dates: First submitted 2018-05-01; First posted 2018-06-06 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomization to intervention or control parallell groups on a 50/50 basis.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study participants were kept blind to treatment allocation by the information that they would be assigned to one of two types of chain blanket, without any information of the difference in weight. The outcome assessor and investigator did not participate in randomization and treatment and were blind to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted metal chain blanket (Experimental): As experimental intervention, a weighted metal chain blanket of 8 kg was used during the night. Using a flexible dose protocol, participants who found the 8 kg blanket too heavy were allowed to change to a 6 kg weighted blanket (see below)
  Interventions: Device: Weighted metal chain blanket
- Control plastic chain blanket (Sham Comparator): As sham comparator, light chain blankets were used, were plastic chains of the same shape and size as the metal chains in the weighted blanket were sewn in. The control blanket has a weight of 1535 grams. When checking the weight of standard blankets for sale in one of the largest stores in Stockholm, weight was ranging from 550 to 2389 grams (average 1332).
  Interventions: Device: Control plastic chain blanket

INTERVENTIONS:
Device: Weighted metal chain blanket — Use of a weighted metal chain blanket of 8 kg
  Arms: Weighted metal chain blanket
Device: Control plastic chain blanket — A blanket with light plastic chains
  Arms: Control plastic chain blanket

SUMMARY:
The aim of the study is to compare an intervention with a weighted metal chain blanket of 8 kg with a control plastic chain blanket of 1,5 kg for patients with Major depressive disorder, bipolar disorder, Generalized Anxiety Disorder (GAD) and/or attention deficit hyperactivity disorder (ADHD) and co-occurring insomnia. Patients are evaluated by a rater blind to treatment allocation with Insomnia Severity Index (ISI), Fatigue Symptom Inventory (FSI), Hospital Anxiety and Depression Scale (HAD) and actigraphy before, during and at primary end-point after 4 weeks use of the blanket.

DETAILED DESCRIPTION:
Insomnia is a common and problematic symptom in many psychiatric disorders. The aim of this study is to evaluate the effect of weighted chain blankets on insomnia and other sleep-related symptoms for patients with Major depressive disorder, Bipolar disorder, Generalized Anxiety Disorder (GAD) and/or ADHD. Potential participants are asked to participate in a study comparing two different types of chain blankets, not mentioning the difference in weight. After signing a informed consent, participants were randomly assigned on a 50/50 basis to a weighted blanket containing metal chains weighing 8 kg or a control blanket containing plastic chains weighing 1,5 kg. Insomnia severity is assessed before and weekly until endpoint at four weeks use of the blanket by a rater blind to treatment allocation. Participants sleep will also be monitored by actigraphy. The controlled phase of the study is followed by a one year open follow up study where all participants are offered to use a weighted blanket of any type.

ELIGIBILITY:
Inclusion Criteria:

• Clinical insomnia for more than two months with a score over 14 points at the Insomnia Severity Index (ISI)1 and a diagnosis of either major depressive disorder, bipolar disorder, Generalized Anxiety disorder (GAD) or ADHD.

Exclusion Criteria:

* active drug abuse,
* overuse of sleep medication,
* illness affecting cognitive functions, such as dementia, schizophrenia, developmental disorders, Parkinson's disease or an acquired brain injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from start to 4 weeks use of the blanket.
  Self-report rating scale assessing the severity of insomnia symptoms. Range 0-28 with higher scores indicating a more severe insomnia

SECONDARY OUTCOMES:
Fatigue Symptom Inventory (FSI) | Change from start to 4 weeks use of the blanket.
  Self-report symptom rating scale for daytime fatigue symptoms. Range 0-130 with higher scores indicating a more severe fatigue.
Actigraphy | Change from start to 4 weeks use of the blanket. .
  An actigraph attached to the arm of the participants on the week before the intervention and during the fourth (last) week of the intervention assessing sleep by interpretation of movement
"Day and night diaries", developed by Assistive technology Stockholm for the evaluation of weighted blankets | Change from start to 4 weeks use of the blanket in patient estimated time (minutes) from going to bed to sleep onset.
  Self reported time to sleep onset.
Hospital Anxiety and Depression Scale (HAD). | Change from start to 4 weeks use of the blanket.
  HAD is a self report rating scale for anxiety and depression symptoms.The HAD is subdivided into subscales for depressive symptoms (HAD-D) and anxiety symptoms (HAD-A), with a range of 0-21 for each subscale. Higher scores indicates more severe symptoms.
Insomnia Severity Index (ISI) | Change from start to 8 weeks, 6 and 12 months use of the blanket
  Self-report rating scale assessing the severity of insomnia symptoms. Range 0-28 with higher scores indicating a more severe insomnia

CONTACTS AND LOCATIONS:
Overall Officials: Mats Adler, M.D. Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Psykiatri Sydväst, Huddinge sjukhus, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ekholm B, Spulber S, Adler M. A randomized controlled study of weighted chain blankets for insomnia in psychiatric disorders. J Clin Sleep Med. 2020 Sep 15;16(9):1567-1577. doi: 10.5664/jcsm.8636. PMID 32536366

DOCUMENTS (1):
  • Study Protocol (2015-11-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT03546036/Prot_000.pdf